CLINICAL TRIAL: NCT00642759
Title: A Phase II Trial of Carboplatin, Abraxane, and Bevacizumab in Previously Untreated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Carboplatin, Abraxane, and Bevacizumab in Previously Untreated Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Suk Heist, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-339
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Abraxane; Carboplatin; Bevacizumab; Avastin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; 130-nm albumin-bound paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Carboplatin, nab-paclitaxel, and bevacizumab
  Interventions: Drug: carboplatin; Drug: Nab-paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: carboplatin — Given by infusion on day 1 of each 3 week cycle for a maximum of 6 cycles
Drug: Nab-paclitaxel — Given by infusion once weekly (days 1, 8 and 15) of each three week cycle for a maximum of 6 cycles
Drug: Bevacizumab — IV infusion

SUMMARY:
The purpose of this research study is to learn more about whether the combination of drugs carboplatin, Abraxane and Avastin helps treat non-small cell lung cancer (NSCLC). One of the standard treatments for advanced NSCLC is the combination of the drugs carboplatin, paclitaxel and Avastin. Paclitaxel can be associated with severe side effects that may make the treatment difficult to tolerate. Some of these side effects are caused by the solution used to dissolve paclitaxel before it can be administered. Abraxane is a different form of paclitaxel that does not need to be dissolved by this solution. Abraxane is approved for the treatment of breast cancer but is not approved to treat NSCLC. We will also be trying to learn more about how the drug Avastin may work to treat cancer.

DETAILED DESCRIPTION:
* Participants will receive a single dose of Avastin 2 weeks before they are scheduled to start the combination of carboplatin, Abraxane and Avastin. Before the dose of Avastin is given, a perfusion CT scan and blood work will be performed. The perfusion CT scan and blood draw will be repeated 12 days after teh Avastin dose (2 days before beginning study treatment).
* The combination of carboplatin, Abraxane and Avastin will be given in 3 week cycles and all drugs will be given as infusions. On day 1, Avastin, Abraxane and carboplatin wil be given. On Day 8 and 15, Abraxane will be given.

Participants can receive up to 6 cycles of carboplatin, Abraxane and Avastin if their disease does not get worse and they do not experience intolerable side effects.

* The following assessment procedures will be performed on day 1 of each cycle: physical exam; routine urine test (every other cycle); Performance status assessment. Routine blood tests will be performed on days 1, 8 and 15.
* Additional procedures performed after cycles 2 and 4 and at 6 months after beginning study treatment are as follows: CT scan, PET scan, perfusion CT and blood work.
* After 6 cycles of carboplatin, Abraxane and Avastin, participants will receive Avastin alone for three weeks. Participants can continue to receive Avastin as long as they do not experience unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-small cell lung carcinoma of non-squamous histology
* AJCC stage IIIB or Stage IV
* Measurable disease by RECIST criteria, and must have at least one target lesion 1cm or greater in diameter for optimal perfusion CT scanning
* No prior chemotherapy treatment or VEGF inhibitor treatment, although prior treatment with EGFR inhibitors will be allowed
* 18 years of age or older
* Adequate bone marrow, renal and liver function as outlined in the protocol

Exclusion Criteria:

* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
* Inadequately controlled hypertension
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke, transient ischemic attack within 6 months prior to study enrollment
* Symptomatic CNS metastases or newly diagnosed CNS metastases that have not yet been definitively treated with radiation and/or surgery. Note that patients with a history of CNS metastases or cord compression are allowed if they have been definitively treated and are clinically stable. Maintenance steroids are allowed. Two weeks need to elapse from the completion of radiation, or 4 weeks from surgery, before starting avastin. Patients do have to remain clinically asymptomatic.
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major medical surgical procedure during the course of the study
* Minor surgical procedure, excluding FNA, core biopsy or placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening
* Pregnant or lactating
* Lung carcinoma of squamous cell histology
* History of hemoptysis within 3 months prior to study enrollment
* Current, on-going treatment with full-dose warfarin or its equivalent at the onset of treatment
* Current or recent (within 10 days of enrollment) use of aspirin or chronic use of other NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Heist, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: carboplatin: Given by infusion on day 1 of each 3 week cycle for a maximum of 6 cycles
  Abraxane: Given by infusion once weekly (days 1, 8 and 15) of each three week cycle for a maximum of 6 cycles
  Bevacizumab
Period: Overall Study
Arm/Group | Chemotherapy
Started | 36
Completed | 35
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression Free Survival Rate
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 36
percentage of participants | 74 [57 to 97]

2. Secondary Outcome: Objective Response Rate to Carboplatin, Abraxane and Avastin
Description: Objective response rate to carboplatin, Abraxane and Avastin according to Response Evaluation Criteria in Solid Tumors [Version 1.0]
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 36
Participants
  Partial Response | 13
  Stable Disease | 13
  Progressive Disease | 2
  Not Evaluable for Response | 8

3. Secondary Outcome: 6 Month Survival Rate
Description: The percentage of participants surviving at least six months after baseline
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants surviving
Arm/Group | Chemotherapy
Number analyzed (Participants) | 36
percentage of participants surviving | 83 [65 to 91]

4. Secondary Outcome: Overall Survival
Description: The median overall survival in months
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy
Number analyzed (Participants) | 36
Months | 13.7 [9.3 to 24.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout duration of study
Description: Adverse events were evaluated on day 1 of cycle 1 and every three weeks prior to chemotherapy and prior to each Avastin dose. Adverse events were then assessed every three months after the completion of 6 cycles of carboplatin, Abraxane, and Avastin until tumor progression or withdrawal from study.
Arm/Group | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 7/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=36)
Thrombosis/thrombus/embolism (Vascular disorders) | 4
Neutrophils (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 1
ALT - SGPT (Metabolism and nutrition disorders) | 1
ALT - SGOT (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=36)
Fatigue (General disorders) | 26
Anorexia (Gastrointestinal disorders) | 10
Dysgeusia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 7
dehydration (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 2
Pain (General disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 15
Neuropathy (Nervous system disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 3
Infection (Infections and infestations) | 4
Renal (Renal and urinary disorders) | 3
Hypertension (Vascular disorders) | 7
Thrombosis/thrombus/embolism (Vascular disorders) | 3
GI bleeding (Gastrointestinal disorders) | 2
Epistaxis (Vascular disorders) | 9
Proteinuria (Metabolism and nutrition disorders) | 3
White Blood Cell Count (Blood and lymphatic system disorders) | 6
Absolute Neutrophil count (Blood and lymphatic system disorders) | 19
Hemoglobin (Blood and lymphatic system disorders) | 20
Platelets (Blood and lymphatic system disorders) | 11
ALT, SGPT (Metabolism and nutrition disorders) | 5
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes